CLINICAL TRIAL: NCT00444067
Title: A Prospective, Multi-Center, Randomized Controlled Study to Compare the Spinal Sealant System as an Adjunct to Sutured Dural Repair With Standard of Care Methods During Spinal Surgery
Brief Title: Study to Evaluate Safety & Effectiveness of Spinal Sealant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DS3-06-002
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2014-09

CONDITIONS: Cerebrospinal Fluid Leakage, Subdural
Keywords: Prevention of CSF leak
MeSH Terms: conditions — Subdural Effusion | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Sealant System (Experimental): Spinal Sealant System
  Interventions: Device: Spinal Sealant
- Standard of Care (Active Comparator): Standard of care methods as an adjunct to sutured dural repair
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Spinal Sealant — Spinal Sealant System
  Arms: Spinal Sealant System
Other: Standard of Care — Standard of Care
  Arms: Standard of Care

SUMMARY:
To evaluate a spinal sealant as an adjunct to sutured dural repair compared to standard of care techniques.

DETAILED DESCRIPTION:
Neurosurgical procedures in the spine often involve incision of the dura mater to access the spinal cord. If the dural incision is not properly repaired and watertight closure is not achieved cerebrospinal fluid (CSF) can escape presenting a risk for significant morbidity. The most frequent complication of CSF leak is recurring headache complicated with symptoms of nausea and vomiting. Furthermore fluid collection under skin prevents proper wound healing and may lead to wound breakdown and infection of the incision or both. Persistent CSF leak has also been associated with the development of cerebellar hemorrhage and subdural hematoma. Primary repair and watertight closure are paramount to minimizing risk and sequelae associated with CSF leak.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for a spinal procedure that requires a dural incision

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jen Doyle, Study Director — Conlfuent Surgical/Covidien
Locations (1):
- Confluent Surgical, Inc., Bedford, Massachusetts, United States

REFERENCES:
- [Derived] Wright NM, Park J, Tew JM, Kim KD, Shaffrey ME, Cheng J, Choudhri H, Krishnaney AA, Graham RS, Mendel E, Simmons N. Spinal sealant system provides better intraoperative watertight closure than standard of care during spinal surgery: a prospective, multicenter, randomized controlled study. Spine (Phila Pa 1976). 2015 Apr 15;40(8):505-13. doi: 10.1097/BRS.0000000000000810. PMID 25646746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was consented on May 15, 2007. The last subject visit occurred on August 12, 2009.
Pre-assignment Details: Washout study, no run-in or wash-out periods.
Groups:
- Spinal Sealant: DuraSeal Spinal Sealant System
- Control: Standard of care methods used as an adjunct to sutured dural repair.
Period: Overall Study
Arm/Group | Spinal Sealant | Control
Started | 74 | 24
Completed | 74 | 23
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Sealant | Control | Total
Number analyzed (Participants) | 74 | 24 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 23 | 92
  >=65 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 9 | 39
  Male | 44 | 15 | 59
Region of Enrollment [Number; unit: participants]
  United States | 74 | 24 | 98
Age (Statistics) [Mean (Standard Deviation); unit: years] | 44.25 (13.06) | 44.70 (11.44) | 44.36 (12.62)

OUTCOME MEASURES:

1. Primary Outcome: Percent(%) Success in Obtaining a Watertight Closure Following Assigned Treatment (Spinal Sealant or Control)
Description: Percent(%) success in obtaining a watertight closure following assigned treatment (Spinal Sealant or Control) where success is defined as:
  A watertight closure of the dural repair intraoperatively after study treatment, confirmed by Valsalva maneuver at 20-25 cm H2O for 5-10 seconds.
Time Frame: Intra-operative
Population: The primary analysis for the primary efficacy endpoint was performed using a two-sided Fisher's Exact Test to test for a difference in the true success rates in obtaining a watertight closure between treatments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Spinal Sealant | Control
Number analyzed (Participants) | 74 | 24
percentage of participants | 98.0 [92.7 to 100] | 79.2 [57.8 to 92.9]

2. Other Pre Specified Outcome: Incidence of Post-Operative CSF Leaks
Description: Percentage of participants with CSF leaks within 90 days post-operatively as determined from clinical diagnosis by one of the following methods:
  * CSF leak or pseudomeningocele related surgical intervention (i.e., breaking skin) within 90 days post-procedure; or
  * CSF leak confirmation by diagnostic testing within 90 days post-procedure; or
  * CSF leak confirmation by clinical evaluation within 90 days post-procedure
Time Frame: 90 Days
Population: Fisher's Exact Test was used to test for a difference in the proportions of subjects with CSF leaks between the two treatments. Confidence intervals were produced based on the observed percentage and also on the percentage estimated using the Kaplan-Meier method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Spinal Sealant | Control
Number analyzed (Participants) | 73 | 24
percentage of participants | 11 [4.9 to 20.5] | 12.5 [2.7 to 32.4]

3. Other Pre Specified Outcome: Incidence of Post-Operative Surgical Site Infections (SSIs)
Description: •Percentage of participants who incur an SSI within 90 days post-procedure determined by clinical diagnosis
  SSIs were diagnosed and classified in accordance with the Centers for Disease Control (CDC) criteria for evaluation and diagnosis of nosocomial surgical site infections and were classified as one of the following (Superficial, Deep or Organ/Space).
Time Frame: 90 Days
Population: Fisher's Exact Test was used to test for a difference in the proportions of subjects with SSIs between the two treatments. Confidence intervals were produced based on the observed percentage and also on the percentage estimated using the Kaplan-Meier method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Spinal Sealant | Control
Number analyzed (Participants) | 73 | 24
percentage of participants | 6.8 [2.9 to 15.7] | 12.5 [4.4 to 35.2]

ADVERSE EVENTS:
Time Frame: 90 Days post-procedure
Arm/Group | Spinal Sealant | Control
Serious Adverse Events (participants affected / at risk) | 17/73 | 5/24
Other Adverse Events (participants affected / at risk) | 64/73 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Sealant (N=73) | Control (N=24)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Incision Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Chemical Meningitis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision Site Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Meningitis Chemical (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrospinal Fistula (Nervous system disorders) | 2 (2) | 2 (2)
Grand Mal Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Loss of Proprioception (Nervous system disorders) | 1 (1) | 0 (0)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Sealant (N=73) | Control (N=24)
Eye Disorders (Eye disorders) | 4 (4) | 3 (3)
Gastrointestinal Disorders (Gastrointestinal disorders) | 11 (11) | 8 (8)
General Disorders and Administration Site Conditions (General disorders) | 19 (19) | 7 (7)
Infections and Infestations (Infections and infestations) | 14 (14) | 7 (7)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 21 (21) | 7 (7)
Investigations (Investigations) | 21 (21) | 7 (7)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 27 (27) | 7 (7)
Nervous System Disorders (Nervous system disorders) | 38 (94) | 13 (34)
Psychiatric Disorders (Psychiatric disorders) | 6 (6) | 2 (2)
Renal and Urinary Disorders (Renal and urinary disorders) | 10 (10) | 6 (6)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Skin and Subcutaneous Disorders (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Vascular Disorders (Vascular disorders) | 9 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* The sponsor can review results at least 30 days prior to public release, and at the request of Sponsor, the PI will withhold submission for an additional period, not to exceed 30 days.
* The first publication of the study results shall be made in conjunction with a joint, multi-center publication of the results. If a multi-center publication is not submitted within 12 months after the conclusion of the study, the PI may publish the results from their individual site.